CLINICAL TRIAL: NCT06012227
Title: Assessment Metabolic Flexibility by Indirect Calorimetry and Circulating Metabolic Parameters in Middle-aged Individuals: The Nutritional Impact of Cheese From Extensive and Intensive Farming.
Brief Title: Assessment Metabolic Flexibility in Middle-aged Individuals: The Nutritional Impact of Cheese Consumption
Acronym: Kent'Erbas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Sebastiano Banni, full professor, University of Cagliari
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UCagliari2
Record Dates: First submitted 2023-07-28; First posted 2023-08-25 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Metabolism; Nutrition
Keywords: metabolic flexibility; lipid metabolism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "kent'erbas" pecorino from extensive farming with crossover Arm 1 (Experimental): This study was a 4-week, randomized, controlled, crossover clinical trial. Arm 1: Volunteers will be randomize to be allocated to eat 350g/week of "kent'erbas" pecorino from extensive farming with a crossover with arm 2 after 6 weeks of washout.
  Interventions: Dietary Supplement: kent'erbas cheese study
- "industrial" pecorino from intensive farming with crossover Arm 2 (Active Comparator): This study was a 4-week, randomized, controlled, crossover clinical trial. Arm 2 : Volunteers will be randomize to be allocated to eat 350g/week of "industrial" pecorino from intensive farming for 4 weeks in total, with a crossover with arm 1 after 6 weeks of washout.
  Interventions: Dietary Supplement: kent'erbas cheese study

INTERVENTIONS:
Dietary Supplement: kent'erbas cheese study — Nutritional intervention with "kent'erbas" pecorino from extensive farming with crossover and "industrial" pecorino from intensive farming

SUMMARY:
The aim of the study will be to evaluate the impact of consumption of meat and dairy products from extensive or intensive farming on apparently healthy individuals aged between 45 and 65 years, a stage of life associated with reduced metabolic flexibility and changes in lipid metabolism.

The study will analyze:

1. The transcription factor PPAR-α determined by the gene expression of PPAR-α in white blood cells, variations in circulating fatty acid metabolism, and the endocannabinoid system determined by circulating analysis of N-acylethanolamine (NAE), and 2-monoacylglycerols (2-MG);
2. Metabolic flexibility, determined by indirect calorimetry in fasting condition during an incremental exercise;
3. Body composition, determined by bioimpedance analysis, waist circumference, and waist-to-hip ratio.

DETAILED DESCRIPTION:
The study will be a double-blind crossover intervention clinical trial conducted on the aforementioned individuals, who will consume "kent'erbas" cheese products, from extensive and intensive farming.

The study will include 105 individuals aged between 45 and 65 years, apparently in good health, recruited from the UTIC cardiology unit of A.O.U.CA Cagliari (Italy). All participants will be provided with a detailed explanation of the study procedures and its purpose, and their participation will be contingent upon signing an informed consent form. Throughout the study, subjects will maintain their regular lifestyle and unrestricted food intake.

At the outset of the study, relevant information necessary for an appropriate approach to each participant will be collected, including a comprehensive medical history, measurement of anthropometric parameters, and blood sampling for a thorough hematological, inflammatory, and lipid-metabolomic analysis.

In the pecorino study, subjects will consume 350g/week of "kent'erbas" pecorino from extensive farming or 350g/week of "industrial" pecorino from intensive farming for 4 weeks in total. At the end of this period, a blood sample will be taken. Subsequently, there will be a 8 weeks washout period during which participants will follow their usual diet without consuming either type of pecorino. At the end of the washout period, an additional blood sample will be taken. Following this, the participants who had consumed "kent'erbas" pecorino will switch to "industrial" pecorino for 4 weeks, and vice versa. At the end of this second period, a final blood sample will be collected.

The quantities of pecorino cheese chosen for intake are representative of the average consumption in Italy.

ELIGIBILITY:
Inclusion Criteria:

* 45-65 years of age
* BMI < 27
* waist-to-hip ratio female<0.85; male < 0.98

Exclusion Criteria:

* metabolic diseases
* Physical activity of competitive nature
* Vegans and vegetarians
* Intolerances and allergies to the foods under study

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 105 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma levels of DHA and acylethanolamides as Metabolic indices of PPAR-α induction increase in plasma levels of DHA | After 4 weeks of treatment, 8 weeks of washout and 4 weeks of crossover
  Changes in plasma levels of DHA)and modulation of the endocannabinoid system, through the biosynthesis of AEA, PEA, and OEA. All these parameters will be assessed as pmoles/ml of plasma

SECONDARY OUTCOMES:
Quotient respiratory changes measurement as metabolic flexibility indices | After 4 weeks of treatment, 8 weeks of washout and 4 weeks of crossover
  Metabolic flexibility indices, through fasting differences in the respiratory quotient, measured as Liter/min of Oxygen consumption and carbon dioxide

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari, Monserrato, Cagliari, Italy